CLINICAL TRIAL: NCT01210677
Title: CArdiac Sarcoidosis Response TO steRoids (CASTOR) Trial
Brief Title: Cardiac Sarcoidosis Response To Steroids Trial
Acronym: CASTOR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding obtained.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, David Birnie, MD, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UOHI-03
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Cardiac Sarcoidosis; Sarcoidosis
Keywords: Cardiac Sarcoidosis; Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone (Active Comparator): Prednisone 0.5 mg/Kg per day orally for 3 months
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Matching placebo tablets(s) taken orally per day
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone 0.5 mg/Kg orally per day for 3 months

SUMMARY:
There are no published clinical consensus guidelines on the treatment of cardiac sarcoidosis. Corticosteroid therapy is advocated by some experts, but is based on small observational studies, with varied clinical response.

Objectives of this trial:

* to systemically assess the response of patients with cardiac sarcoidosis, to treatment with corticosteroids
* to identify the clinical predictors of response to treatment with corticosteroids
* to assess the utility of imaging with PET and MRI to predict response to treatment with corticosteroids
* to determine the prevalence of cardiac sarcoidosis in young patients with unexplained heart block and in patients with unexplained dilated cardiomyopathy associated with ventricular tachycardia
* to use the data from this pilot study to assess the need, feasibility, and sample size for a larger multicentre trial

ELIGIBILITY:
Inclusion Criteria:

* evidence of clinical cardiac sarcoidosis causing significant conduction system disease (defined as complete right bundle branch block and left axis deviation or left bundle branch block or second or third degree AV block in young patients (< 60 yrs) AND/OR
* evidence of clinical cardiac sarcoidosis causing non-ischemic dilated cardiomyopathy and sustained ventricular tachycardia AND
* PET or MRI imaging supporting the diagnosis of cardiac sarcoidosis

Exclusion Criteria:

* unable or unwilling to provide informed consent
* history of noncompliance of medical therapy
* patients with active infection
* patients with active inflammatory disease not related to sarcoidosis
* patients with other known causes of heart block or LV dysfunction
* patients with known active malignancy
* patients wwho are pregnant or lactating
* patients with other indications for steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Heart failure hospitalization and sustained ventricular arrhythmia | 3 months
  Considered a responder to steroid therapy if alive, no heart failure hospitalization and no sustained ventricular arrhythmia, and improvement in one or both of:
  1. LV function (defined as 5% increase in EF units or 10% decrease in volumes)
  2. greater than or equal to one heart block grade (defined as improvement from eg. third to second degree AV block or resolution of bundle branch block)

SECONDARY OUTCOMES:
Change in disease activity by PET imaging | 3 months
  1. Change in disease activity as assessed by PET imaging (comparing pre-treatment to 3 month scans)
  2. Atrial fibrillation burden during the 3 month treatment period (from pacemaker or ICD diagnostics)
  3. Ventricular arrhythmia burden during the 3 month treatment period
  4. Percent of ventricular pacing (pacemaker programming will be standardized in all patients)
  5. Patient Quality of life (using SF-36 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: David Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Pablo B. Nery, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada